CLINICAL TRIAL: NCT05173194
Title: Effects of a Remotely Supervised Exercise Program on Inflammatory Markers, Muscle Strength and Lung Function in Adult Patients With Cystic Fibrosis
Brief Title: Remotely Supervised Exercise for Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Margarita Perez, Professor in Exercise Physiology, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FQKloE-II
Record Dates: First submitted 2021-11-23; First posted 2021-12-29 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Exercise program; Lung funcion; Inflammation
MeSH Terms: conditions — Cystic Fibrosis; Inflammation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Evaluators of outcomes will be masked as for the study group of each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telematic Exercise (Experimental): A remotely supervised resistance exercise program will be carried out for 8 weeks, with three weekly sessions lasting approximately 60 minutes each. Training will be performed in groups of four patients, according to their lung function/physical fitness. The first training session will be on site (University) for familiarization, planning and adjustment of the exercises, and the following sessions will be performed online. Each session is divided into: (i) Warm-up and joint mobility; (ii) main part: strength exercises for different muscle groups; and (iii) cool down: stretching and breathing exercises.
  Interventions: Other: Exercise
- Control (No Intervention): Control group will follow routine recommendations from the multidisciplinary CF team.

INTERVENTIONS:
Other: Exercise — Eight-week program of a remotely supervised resistance exercise. Frequency: three times per week. Duration: 60 minutes per session. Training program: warm-up and joint mobility; strength exercises for different muscle groups; and cool down (stretching and breathing exercises).
  Arms: Telematic Exercise

SUMMARY:
Cystic fibrosis (CF) is a genetic disease characterized by abnormal chloride transport in epithelial tissues. Inflammation is a key component contributing to the main alterations induced by the disease. The increase in life expectancy comes with a higher prevalence of CF-related comorbidities, but also with new emerging complications directly related to aging. Physical fitness and exercise practice have been previously associated to survival and better quality of life in patients with cystic fibrosis. Thus, the aim of this study is to assess the effects of a remotely supervised resistance exercise program on lung function, muscle strength, body composition, quality of life and inflammatory markers in adult patients with cystic fibrosis.

DETAILED DESCRIPTION:
This study aims to assess the effects of a remotely supervised resistance exercise program on lung function, muscle strength, body composition, quality of life and inflammatory markers in adult patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed clinical and genetic diagnosis for cystic fibrosis;
* Age from 16 years.

Exclusion Criteria:

* Musculoskeletal disorders that do not allow the performance of physical exercise;
* Pregnancy;
* Absence of registration of clinical required.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Change in peripheral muscle strength. Upper and lower limb muscle strength will be evaluated using the 5 maximum repetition test in specific strength machines. Handgrip strength will be measured with a dynamometer. | Baseline and 8 weeks
  Change from baseline to 8 weeks
Change in body composition (muscle mass and skeletal mass index - kg/m2) measured through dual-energy x-ray absorptiometry (DEXA) | Baseline and 8 weeks
  Change from baseline to 8 weeks
Change in plasmatic levels of Klotho | Baseline and 8 weeks
  Change from baseline to 8 weeks
Change in plasmatic levels of interleukins (IL-8 and IL-10) | Baseline and 8 weeks
  Change from baseline to 8 weeks

SECONDARY OUTCOMES:
Change in Pulmonary Function (Lung Function) | Baseline and 8 weeks
  Change from baseline to 8 weeks
Change in quality of life evaluated using the Cystic Fibrosis Questionnaire (CFQ-R +14). Scores range from 0 to 100 with higher scores corresponding to better quality of life. | Baseline and 8 weeks
  Change from baseline to 8 weeks
Change in inspiratory muscle strength (MIP) | Baseline and 8 weeks
  Change from baseline to 8 weeks
Change in functional capacity (30 seconds sit-to-stand test) | Baseline and 8 weeks
  Change from baseline to 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Margarita Perez-Ruiz, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Hospital La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van de Weert-van Leeuwen PB, Hulzebos HJ, Werkman MS, Michel S, Vijftigschild LA, van Meegen MA, van der Ent CK, Beekman JM, Arets HG. Chronic inflammation and infection associate with a lower exercise training response in cystic fibrosis adolescents. Respir Med. 2014 Mar;108(3):445-52. doi: 10.1016/j.rmed.2013.08.012. Epub 2013 Aug 28. PMID 24480322
- [Background] Vendrusculo FM, Heinzmann-Filho JP, da Silva JS, Perez Ruiz M, Donadio MVF. Peak Oxygen Uptake and Mortality in Cystic Fibrosis: Systematic Review and Meta-Analysis. Respir Care. 2019 Jan;64(1):91-98. doi: 10.4187/respcare.06185. Epub 2018 Sep 11. PMID 30206131
- [Background] Vandekerckhove K, Keyzer M, Cornette J, Coomans I, Pyl F, De Baets F, Schelstraete P, Haerynck F, De Wolf D, Van Daele S, Boone J. Exercise performance and quality of life in children with cystic fibrosis and mildly impaired lung function: relation with antibiotic treatments and hospitalization. Eur J Pediatr. 2017 Dec;176(12):1689-1696. doi: 10.1007/s00431-017-3024-7. Epub 2017 Sep 30. PMID 28965267
- [Background] Perez M, Groeneveld IF, Santana-Sosa E, Fiuza-Luces C, Gonzalez-Saiz L, Villa-Asensi JR, Lopez-Mojares LM, Rubio M, Lucia A. Aerobic fitness is associated with lower risk of hospitalization in children with cystic fibrosis. Pediatr Pulmonol. 2014 Jul;49(7):641-9. doi: 10.1002/ppul.22878. Epub 2013 Sep 9. PMID 24019231
- [Background] Mostafidi E, Moeen A, Nasri H, Ghorbani Hagjo A, Ardalan M. Serum Klotho Levels in Trained Athletes. Nephrourol Mon. 2016 Jan 9;8(1):e30245. doi: 10.5812/numonthly.30245. eCollection 2016 Jan. PMID 26981496
- [Background] Gao W, Yuan C, Zhang J, Li L, Yu L, Wiegman CH, Barnes PJ, Adcock IM, Huang M, Yao X. Klotho expression is reduced in COPD airway epithelial cells: effects on inflammation and oxidant injury. Clin Sci (Lond). 2015 Dec;129(12):1011-23. doi: 10.1042/CS20150273. Epub 2015 Jul 10. PMID 26201096
- [Background] Kureya Y, Kanazawa H, Ijiri N, Tochino Y, Watanabe T, Asai K, Hirata K. Down-Regulation of Soluble alpha-Klotho is Associated with Reduction in Serum Irisin Levels in Chronic Obstructive Pulmonary Disease. Lung. 2016 Jun;194(3):345-51. doi: 10.1007/s00408-016-9870-7. Epub 2016 May 2. PMID 27140192
- [Background] Krick S, Baumlin N, Aller SP, Aguiar C, Grabner A, Sailland J, Mendes E, Schmid A, Qi L, David NV, Geraghty P, King G, Birket SE, Rowe SM, Faul C, Salathe M. Klotho Inhibits Interleukin-8 Secretion from Cystic Fibrosis Airway Epithelia. Sci Rep. 2017 Oct 30;7(1):14388. doi: 10.1038/s41598-017-14811-0. PMID 29085059
- [Background] Amaro-Gahete FJ, de-la-O A, Jurado-Fasoli L, Gutierrez A, Ruiz JR, Castillo MJ. Association of physical activity and fitness with S-Klotho plasma levels in middle-aged sedentary adults: The FIT-AGEING study. Maturitas. 2019 May;123:25-31. doi: 10.1016/j.maturitas.2019.02.001. Epub 2019 Feb 5. PMID 31027673
- [Background] Amaro-Gahete FJ, De-la-O A, Jurado-Fasoli L, Espuch-Oliver A, de Haro T, Gutierrez A, Ruiz JR, Castillo MJ. Exercise training increases the S-Klotho plasma levels in sedentary middle-aged adults: A randomised controlled trial. The FIT-AGEING study. J Sports Sci. 2019 Oct;37(19):2175-2183. doi: 10.1080/02640414.2019.1626048. Epub 2019 Jun 4. PMID 31164040
- [Background] Amaro-Gahete FJ, De-la-O A, Jurado-Fasoli L, Espuch-Oliver A, Robles-Gonzalez L, Navarro-Lomas G, de Haro T, Femia P, Castillo MJ, Gutierrez A. Exercise training as S-Klotho protein stimulator in sedentary healthy adults: Rationale, design, and methodology. Contemp Clin Trials Commun. 2018 May 18;11:10-19. doi: 10.1016/j.conctc.2018.05.013. eCollection 2018 Sep. PMID 30023455
- [Background] Kriemler S, Kieser S, Junge S, Ballmann M, Hebestreit A, Schindler C, Stussi C, Hebestreit H. Effect of supervised training on FEV1 in cystic fibrosis: a randomised controlled trial. J Cyst Fibros. 2013 Dec;12(6):714-20. doi: 10.1016/j.jcf.2013.03.003. Epub 2013 Apr 13. PMID 23588193
- [Background] Rovedder PM, Flores J, Ziegler B, Casarotto F, Jaques P, Barreto SS, Dalcin Pde T. Exercise programme in patients with cystic fibrosis: a randomized controlled trial. Respir Med. 2014 Aug;108(8):1134-40. doi: 10.1016/j.rmed.2014.04.022. Epub 2014 Jun 26. PMID 25002195